CLINICAL TRIAL: NCT07091591
Title: "Why do the Recommendations Keep Changing?" A Randomized Controlled Trial of a Scrollytelling Web Application to Help Members of the Public Understand Better How and Why Public Health Guidelines Change Over Time
Acronym: Changing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Holly Witteman, Professor, Dr. Holly witteman, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Changing; VR5-172668 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Social Perception; Psychology
Keywords: Public Health Agency of Canada; Public health guidelines; Scientific skepticism; Nutrition; Food policy; Nutrition guidelines

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: We will use computerized randomization within Qualtrics to automatically assign participants to study arms randomly. We will use masking in R statistical software to blind analysts/investigators to the group assignment of each participant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pandemic (Experimental): Web page explaining the reasons for shifting recommendations in the context of a pandemic.
  Interventions: Behavioral: Changing (version: pandemic)
- Nutrition (Active Comparator): Web page explaining the reasons for shifting recommendations in the context of nutrition.
  Interventions: Behavioral: Changing (version: nutrition)
- Control (No Intervention): No material of information is provided

INTERVENTIONS:
Behavioral: Changing (version: pandemic) — The application explains that, faced with a complex situation such as a pandemic, decision-makers have to navigate through uncertainty, often without knowing exactly how the situation will evolve. Scientific research guides their choices, but early studies can sometimes prove inaccurate and require adjustments. For example, during the COVID-19 pandemic, some initial studies showed that certain drugs could help, but more rigorous research showed that they were not effective. Over time, accumulated knowledge enables us to better understand the situation and make informed decisions. Lessons learned from past crises help to better prepare for future complex situations.
  Arms: Pandemic
Behavioral: Changing (version: nutrition) — The intervention discusses the evolving nature of scientific research on diet and health. It explains how initial studies can suggest one thing, only for later studies to offer new insights or clarify previous findings. For example, while early research linked high fat intake with heart disease, more recent studies have shown that some fats, like those in nuts, avocados, and oily fish, are actually beneficial. It emphasizes that science often advances gradually, and rigorous, long-term studies help understanding. It also points out that health recommendations are influenced by multiple factors, and over time, accumulated knowledge enables us to better understand the situation and make informed decisions.
  Arms: Nutrition

SUMMARY:
This study will be an online 3-arm randomized controlled trial. Here intervention group 1 will receive the intervention in the form of an animated cartoon "scrollytelling" outlining the various changes and reasons for changes in public health guidelines in the context of nutrition (e.g. recommendations on fat intake). Intervention group 2 will have a scrollytelling on the reasons why public health recommendations always change in the context of infectious disease control (e.g. during the COVID-19 pandemic). And finally, the control group will receive no intervention.

DETAILED DESCRIPTION:
The project was initially conceived on Figma, a design platform, enabling our design team to create a user interface. Following this design phase, our experienced developers took over, using the Vue.js framework. Development involved fundamental web languages: JavaScript, CSS and HTML. JavaScript made the interface dynamic for smooth user interaction, CSS applied the detailed visual design conceived on Figma, and HTML structured the application's content. This combination resulted in an application, showcasing Vue.js's effectiveness in application development. Our intervention was the "Changing" application, which was a scrollytelling that, in its two versions (food and pandemic), explained why and how public health guidelines are being changed. The main purpose of the "Changing" application is to explain the reasons for ongoing changes in public health guidelines, using COVID-19 and nutrition as examples.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit participants who are aged 18 years or older. They will be able to provide written informed consent, and be able to read and understand French or English. Additionally, they should be able to use a computer.

Exclusion Criteria:

* We will exclude participants who are younger than 18 years old, unable to provide written informed consent, unable to read or understand French or English, or unable to use a computer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Anti-intellectualism | Immediately after intervention
  Anti-intellectualism can be defined as "the refusal to recognize the pre-eminence of intelligence and the value of the sciences". Richard Hofstadter (1963) described anti-intellectualism generally as " a resentment and distrust of the things of the mind and those who represent it" (Hofstadter 1966). This sentiment is captured through a set of six items measuring attitudes towards various authoritative figures and institutions, including medical doctors, scientists, economists , teachers, expert and the Public Health Agency of Canada (Merkley and Loewen 2021). These attitudes are typically assessed using a Likert scale, a widely used semantic rating system in surveys that offers respondents a nuanced range of responses (typically 5 or 7 options) to gauge their perceptions, attitudes, and opinions accurately. Unlike binary "Yes" or "No" responses, this scale allows for a more detailed understanding of how individuals perceive and intercept the issues under investigation.

SECONDARY OUTCOMES:
Knowledge-changing | Immediately after intervention
  This variable measured individuals perceptions and beliefs concerning various aspects of scientific knowledge and its role in public health decisions. Items addressed the relationship between scientific discoveries, political decisions and the evolution of knowledge.
  It is a discrete quantitative variable whose score ranges from 0 to 10, with the answers to the ten questions being true=1 or false=0.

CONTACTS AND LOCATIONS:
Locations (1):
- Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
We will make anonymized data available on Boréalis, Université Laval's Dataverse.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: As soon as the manuscript describing the results is posted as a preprint.
Access Criteria: No restrictions.